CLINICAL TRIAL: NCT07155538
Title: Validity and Reliability of the Bed Bridge Test in Acute Stroke Patients
Brief Title: Bed Bridge Test in Acute Stroke Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Gaziantep Islam Science and Technology University (Other)
Responsible Party: Principal Investigator, Zekiye İpek, Assoc.Prof., Gaziantep Islam Science and Technology University
Other Study IDs: ipekkirmaci...
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Stroke, Acute
Keywords: stroke; validity; reliability; bed bridge test
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assesment test for Validity and Reliability — Assesment test

SUMMARY:
Studies examining the validity and reliability of easy-to-apply muscle strength and mobility outcome measures in the acute and subacute phases of stroke are quite limited. Therefore, the purpose of this study was to investigate whether the In-Bed Bridge Test is a useful outcome measure for assessing lower extremity muscle strength and mobility in stroke.

DETAILED DESCRIPTION:
Stroke is defined as an acute neurological dysfunction of vascular origin, with symptoms varying depending on the affected brain regions. Stroke patients often experience spasticity, upper and lower extremity dysfunction, mobility loss, and problems with walking, swallowing, vision, and communication, which span multiple systems and impact an individual's functionality. Assessing functional mobility and muscle strength plays a crucial role in planning a stroke patient's treatment program and demonstrating treatment effectiveness. Studies examining the validity and reliability of easily administered muscle strength and mobility outcome measures in the acute and subacute stages of stroke are relatively few. Therefore, the purpose of this study was to investigate whether the In-Bed Bridge Test is a useful outcome measure for assessing lower extremity muscle strength and mobility in stroke.

ELIGIBILITY:
Inclusion Criteria:

* medically stable
* ischemic or hemorrhagic stroke within six months.
* 40 years of age or older,
* have no other known neurological or orthopedic problems,
* have a Mini Mental Test score of 24 or higher.

Exclusion Criteria:

-diagnosed with cognitive impairment and those with communication and cooperation problems

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute Stroke Patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-25 (Estimated)

PRIMARY OUTCOMES:
Bed Bridge Test | At baseline and second day
  The bed bridge test is performed on a bed or stretcher with a zero-degree headrest. The upper extremity is extended parallel to the trunk. The knees and hips are flexed at 45° and 60°, respectively, and measured and controlled with a goniometer. The in-bed bridge test is performed in four different ways: two with a limited number of repetitions (5 and 10) and two with a time limit (30 and 60 s). For the 5 and 10 repetitions limited versions of the in-bed bridge, participants are asked to perform 5 and 10 repetitions as quickly as possible, and the time required to complete each repetition is recorded. For the time-limited version of the bed bridge pose, participants are asked to complete as many repetitions as possible within 30 and 60 seconds, and the number of repetitions is recorded.
Short Physical Performance Battery Test | At baseline
  It consists of three objective tests that assess lower body function. These are: the 4-meter walk test, the chair-to-stand test, and the standing balance test. A 5-level summary score (0-4) is assigned to each test. A score of zero indicates "Unable to perform." Participants included in the "Unable to perform" category were:
  1. Those who attempted but were unable to perform the activity,
  2. The interviewer or the subject felt unsafe,
  3. Those unable to perform the activity due to other health reasons.
The National Institutes of Health Stroke Scale (NIHSS) | At baseline
  The National Institutes of Health Stroke Scale (NIHSS), consisting of 11 basic scales based on physical examination findings, was developed to determine stroke severity. This scoring system provides insight into patient prognosis and response to treatment.An increase in the score indicates an increase in stroke severity.
Fugl-Meyer Rating Scale | At baseline
  The Fugl-Meyer Rating Scale (FMRS) will be used to assess lower extremity motor function. This scale was developed to assess a patient's sensorimotor recovery after stroke according to the Brunnstrom stages of motor recovery. It consists of five sections: motor function (upper and lower extremities), sensation, balance, range of motion, and joint pain. In our study, the lower extremity assessment section will be used. The total possible score for the lower extremity is 34. The higher the score, the better the performance. Each parameter is scored as 0: Failure, 1: Partially Successful, and 2: Completely Successful.
Sit-to-Stand Test | At baseline
  This test is used to assess the patient's functional status. The participant is asked to sit with their feet flat on a standard chair, 43-46 cm high, with no armrests and a backrest. The participant is asked to stand up from the chair and sit down again for one minute, arms crossed in front of the chest. The total number of sit-ups completed constitutes the total score.